CLINICAL TRIAL: NCT00457210
Title: The Influence of the Radiotherapy or Stereotactic Radiosurgery on the Cognitive Function of the Patients With the Neurotrax Assessment System and a Cognitive Questionnaire.
Brief Title: The Influence of Radiotherapy on Cognitive Function
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Mindstreams (Unknown)
Other Study IDs: TASMC-07-BC-040-CTIL
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Last update posted 2007-04-06 (Estimated); Status verified 2007-04

CONDITIONS: Radiotherapy; Brain Neoplasms; Quality of Life
Keywords: Psychology
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

INTERVENTIONS:
Procedure: Brain Radiotherapy/Stereotactic Radiosurgery

SUMMARY:
The cognitive function of 150 patients that undergone any Radiotherapy treatment to the brain will be assessed at 3 time points before and after the treatment.

DETAILED DESCRIPTION:
The basic cognitive function and QOL of 150 oncologic patients that undergone Radiotherapy or Radiosurgery treatment to the brain due to primary tumor, metastases or increased risk of brain metastases, will be assessed at 3 time points: before the treatment, immediately after the treatment, and on the next follow up visit. The assessment tools that will be used are Neurotrax standard cognitive computerized tests and 2 short questionnaires.Patients that will receive a one-day treatment will be tested on 2 time points only- before the treatment and on FU.The research will reveal the positive and the negative influences of the Radiotherapy, along with the assessment of norms for the cognitive function and quality of life of oncologic patients being treated by RT.Eligibility criteria:oncologic patients of both genders, with primary brain tumors, metastases or with increased risk of brain metastases, that are referred to conformal/palliative or preventive Radiotherapy treatment or to Stereotactic Radiosurgery, who are able to follow instructions in Hebrew.The participants will be 20-80 years old.Main comparisons will be performed between the cognitive tests results on 3 time points mentioned. The study will continue until the needed number of participants will be achieved.

ELIGIBILITY:
Inclusion Criteria:

* 20-80 years old oncologic patients, of both genders, that are referred to Brain Radiotherapy or Stereotactic Radiosurgery due to primary brain tumor/ brain metastases or increased risk for brain metastases.
* Are able to follow instructions in Hebrew.

Exclusion Criteria:

* Non-Hebrew speakers can not participate.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2007-04

CONTACTS AND LOCATIONS:
Overall Officials: Ben Corn, PhD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv sourasky Medical Center, Tel Aviv, Israel